CLINICAL TRIAL: NCT05597280
Title: Bedaquiline Enhanced Post ExpOsure Prophylaxis for Leprosy: Phase 3 Study
Brief Title: Bedaquiline Enhanced Post ExpOsure Prophylaxis for Leprosy
Acronym: BE-PEOPLE P3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BE-PEOPLE Phase 3
Record Dates: First submitted 2022-10-03; First posted 2022-10-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE-PEP (Experimental): Intervention arm in which BE-PEP will be provided to all persons residing within 100 meters of an index case, to be repeated after four weeks for household contacts.
  BE-PEP: bedaquiline (400 or 800 mg depending on weight band) combined with rifampicin (10 mg/kg) will be provided as post-exposure prophylaxis
  Both arms will target anyone living within 100 meters of an index case or the entire village if more than 50% are eligible. The dosage form of rifampicine is 150 mg and 300 mg, for bedaquiline it's 20 mg or 100 mg.
  Interventions: Drug: BE-PEP Bedaquiline; Drug: BE-PEP Rifampicin
- SDR PEP (Active Comparator): WHO recommended standard PEP will be provided, i.e. 10 mg/kg of rifampicin in a single dose. In both arms anyone living within 100 meters of an index case will be targeted or the entire village if more than 50% are eligible.
  The dosage form of rifampicine is 150 mg and 300 mg.
  Interventions: Drug: SDR-PEP Rifampicin

INTERVENTIONS:
Drug: BE-PEP Bedaquiline — bedaquiline
  Arms: BE-PEP
Drug: SDR-PEP Rifampicin — SDR-PEP: rifampicin
  Arms: SDR PEP
Drug: BE-PEP Rifampicin — BE-PEP rifampicin
  Arms: BE-PEP

SUMMARY:
There will be two study arms. Arm 1 will be the intervention arm in which there will be provided BE-PEP to all persons residing within 100 meters of an index case, to be repeated after four weeks for household contacts. Arm 2 will be the comparator arm in which the WHO recommended standard PEP will be provided, i.e. 10 mg/kg of rifampicin in a single dose. In both arms the investigators will target anyone living within 100 meters of an index case or the entire village if more than 50% are eligible. Provision of BE-PEP will start in 2023 and follow-up will continue until 2026. The main study outcome will be the comparison of leprosy risk in individuals that received BE-PEOPLE standard WHO SDR-PEP versus individuals that received BE-PEP. In addition the investigators will compare the overall leprosy incidence over the follow-up period between the two study arms.

DETAILED DESCRIPTION:
Assuming the phase 2 study will not reveal any drug related adverse events and following the advice of the DSMB and the involved ethics committees, the investigators will proceed with a phase 3 study for which randomization will take place in December, 2022. There will be two study arms. Arm 1 will be the intervention arm in which there will be provided BE-PEP to all persons residing within 100 meters of an index case, to be repeated after four weeks for household contacts. Arm 2 will be the comparator arm in which the WHO recommended standard PEP will be provided, i.e. 10 mg/kg of rifampicin in a single dose. In both arms anyone living within 100 meters of an index case will be targeted or the entire village if more than 50% are eligible. Provision of BE-PEP will start in 2023 and follow-up will continue until 2026. The main study outcome will be the comparison of leprosy risk in individuals that received standard WHO SDR-PEP versus individuals that received BE-PEP. In addition the overall leprosy incidence over the follow-up period will be compared between the two study arms. As stated above, the primary outcome measure will be the incidence rate ratio of leprosy between those who received BE-PEP and those who received the standard SDR-PEP. From this analysis the investigators will exclude those not eligible for BE-PEP, i.e. children below 5 years of age and/or with a weight below 20 kg. A Poisson model will be fit with village nested in island as random effect and controlled for distance to the nearest index case at baseline. In addition the investigators will compute incidence rate ratios between the entire BE-PEP and SDR-PEP arms over the period 2023-2026, also based on a Poisson model with village nested in island as random effect. Throughout the BE-PEOPLE trial the investigators will continue sampling leprosy patients identified (a skin biopsy from the edge of non-facial lesions), with the aim of using molecular assays for M. leprae as quality assurance mechanism. If sufficient DNA is available Deeplex-MycLep will be used for typing the strains, which will allow to perform highly sensitive surveillance for (traces of) resistance to rifampicin and bedaquiline. As part of BE-PEOPLE, the investigators will moreover enroll all microbiologically confirmed tuberculosis patients on all islands of Comoros (Moheli, Anjouan, and Grande Comore, where bedaquiline will not be introduced, maximum 100 patients/ year) and assess whether they ever received (BE-)PEP or leprosy treatment. The investigators will genotype their sputum with Deeplex-MycTB XL, which includes all M. tuberculosis genes (potentially) involved in resistance to rifampicin and bedaquiline, to be able to detect the earliest traces of acquired resistance to these drugs, which is unexpected after single dose administration.The overall goal of BE-PEOPLE is to validate a robust and safe leprosy PEP regimen, and its optimal administration, that prevents leprosy in the individual and interrupts transmission at the village level.If BE-PEP turns out to be safe and successful, the investigators aim to adjust national guidelines in Comoros towards island wide implementation on Anjouan and Moheli, allowing to sustainably eliminate leprosy.

ELIGIBILITY:
Inclusion Criteria:

1. Living in one of the study clusters (34 on Anjouan, 10 on Mohéli), in good state of health
2. Aged 2 years and above, as leprosy is very rare among infants and young toddlers. Children age 2-4 years or weighing less than 20 kg will not be given bedaquiline. If eligible they will receive only rifampicin.
3. Able and willing to provide informed consent for leprosy and tuberculosis screening, and PEP administration (as applicable in the different arms)

Exclusion Criteria:

1. Signs of active leprosy
2. Signs of active pulmonary tuberculosis (cough ≥2 weeks duration and without a negative TB test)
3. Signs of active extra-pulmonary tuberculosis (bluish-red nodules that cover the lymph nodes, bones or joints, or cervical glands with discharge)
4. Having received rifampicin or bedaquiline (if applicable) in the last 2-year period
5. Self-reported (suspected) pregnancy or breastfeeding
6. Concurrent (within the last three week period before D0) use of medications not included in the safe list (for bedaquiline only)

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 124000 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate effectiveness of PEP based on a combination of rifampicin and bedaquiline (BE-PEP), in preventing leprosy among contacts of incident cases. | Through study completion, an average of 4 years
  The incidence rate ratio of leprosy between contacts who received the trial regimen (BE-PEP: rifampicin 600 mg plus bedaquiline 800mg, repeated once after four weeks for household contacts) and those who received the WHO standard prophylactic regimen (SDR-PEP: rifampicin 600 mg, single dose).

SECONDARY OUTCOMES:
To assess effectiveness of the BE-PEP regimen at village level. | Through study completion, an average of 4 years
  The incidence rate ratio between villages that received BE-PEP and villages that received SDR-PEP.
To quantify frequency of potential adverse events such as gastro-intestinal (nausea, vomiting), nervous system-related (headache, dizziness) and cutaneous reactions | Until day 30 after treatment administration. 2026 final analyses
  The proportion of participants treated with BE-PEP that report adverse events, with a breakdown by type of event.
To assess anti-PGL-I sero surveys as a tool to monitor leprosy transmission | Through study completion, an average of 4 years
  anti-PGL-I sero prevalence rates in villages belonging to arm 4 of the original PEOPLE trial at the time of the first survey round in 2019 and the final round of BE-PEOPLE in 2026
To monitor rifampicin and bedaquiline resistance among leprosy and tuberculosis patients | Through study completion, an average of 4 years
  The investigators will quantify the prevalence of rifampicin and/or bedaquiline resistant strains of M. leprae and M. tuberculosis on each of the study islands making use of molecular markers.
To assess cost-effectiveness of the BE-PEP regimen compared to SDR-PEP. | Through study completion, an average of 4 years
  Cost per case averted between BE-PEP arm and SDR-PEP.
To evaluate the viability of Mycobacterium tuberculosis during and after treatment among TB patients on Grande Comore. | Through study completion, an average of 4 years
  The change in viability of Mycobacterium tuberculosis in subsequent samples of TB patient undergoing treatment on Grande Comore

CONTACTS AND LOCATIONS:
Overall Officials: Younoussa Assoumani, Principal Investigator — Damien Foundation Comoros
Locations (1):
- Fondation Damien, Moroni, Comoros

REFERENCES:
- [Derived] Younoussa A, Samidine SN, Bergeman AT, Piubello A, Attoumani N, Grillone SH, Braet SM, Tsoumanis A, Baco A, Mzembaba A, Salim Z, Amidy M, Grillone S, Snijders R, Corstjens P, Ortuno-Gutierrez N, Hoof C, Geluk A, de Jong BC, Hasker E. Protocol, rationale and design of BE-PEOPLE (Bedaquiline enhanced exposure prophylaxis for LEprosy in the Comoros): a cluster randomized trial on effectiveness of rifampicin and bedaquiline as post-exposure prophylaxis of leprosy contacts. BMC Infect Dis. 2023 May 9;23(1):310. doi: 10.1186/s12879-023-08290-0. PMID 37161571